CLINICAL TRIAL: NCT02325570
Title: The Evaluation of the Clinical Effects of the KLOX BioPhotonic OraLum Gel With a LED Curing Lamp as an Adjunct to the Non-Surgical Treatment of Moderate to Severe Chronic Periodontitis
Brief Title: Evaluation of the KLOX BioPhotonic OraLum Gel With a LED Curing Lamp in Moderate to Severe Chronic Periodontitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KLOX Technologies Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CL-K1004-P001
Record Dates: First submitted 2014-12-17; First posted 2014-12-25 (Estimated); Last update posted 2016-02-23 (Estimated); Status verified 2016-02

CONDITIONS: Moderate to Severe Chronic Periodontitis
MeSH Terms: interventions — Tooth Exfoliation; Root Planing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- KLOX BioPhotonic OraLum Gel + SRP (Experimental): Split-mouth design:the half-mouth randomly selected will be treated with KLOX BioPhotonic OraLum gel (with a LED curing lamp) as an adjunct to SRP.
  Interventions: Device: KLOX BioPhotonic OraLum Gel; Procedure: Scaling and Root Planing (SRP)
- Scaling and Root Planing (SRP) (Other): The second half-mouth will be treated with SRP alone.
  Interventions: Procedure: Scaling and Root Planing (SRP)

INTERVENTIONS:
Device: KLOX BioPhotonic OraLum Gel — Klox BioPhotonic OraLum Gel will be used with a LED curing lamp as an adjunct to conventional non-surgical periodontal treatment (SRP).
  Arms: KLOX BioPhotonic OraLum Gel + SRP
Procedure: Scaling and Root Planing (SRP) — Scaling and Root Planing (SRP) is the conventional non-surgical treatment of chronic periodontitis.

SUMMARY:
Multicenter, prospective, interventional open case series study using a randomized split-mouth design in moderate to severe chronic periodontitis patients having half-mouth treated with the KLOX BioPhotonic OraLum gel with a LED curing lamp as an adjunct to conventional non-surgical periodontal treatment (SRP) versus SRP alone in the second (control) half-mouth.

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated written informed consent form;
2. Male or female patients aged 18 years old and above;
3. Good general health, free of systemic diseases such as diabetes, arthritis, HIV infection or genetic disorder that could influence the outcome of the treatment;
4. Patient with clinically confirmed signs and symptoms of generalized moderate to severe chronic periodontitis (as defined according to International Classification of Periodontal Diseases, Armitage 1999);
5. Patient has had no periodontal treatment for the last year prior to the study;
6. Females of childbearing potential must not be pregnant nor lactating at study entry and agree to use an adequate contraceptive method during the study.

   Inclusion Criteria Post Oral Hygiene Instructions (OHI):
7. Patient demonstrates sufficient plaque control as indicated by a plaque score < 30% after hygiene period;
8. Patient has at least two sites in each quadrant with probing pocket depth (PPD) equal or more than 5 mm or equal or less than 7 mm.

Exclusion Criteria:

1. Patient with an existing aggressive periodontitis;
2. Presence of oral local mechanical factor(s) that could, in the opinion of the investigator, influence the outcome of the study;
3. Presence of orthodontic appliances, or any removable appliances, that impinges on the tissues being assessed;
4. Soft or hard tissue tumours of the oral cavity;
5. Systemic antibiotic therapy or anti-inflammatory drugs or any other medication(s) that might interfere with periodontal healing within the last three months prior to study entry and throughout the study duration;
6. Patient has participated in any other clinical study within 30 days prior to study entry and throughout the study duration;
7. Use of anticoagulants such as warfarin, clopidogrel, enoxaparin or high doses of aspirin (162 mg daily);
8. Regular use of chlorhexidine oral rinses / mouthwashes (Non-medicated, over the counter, mouthwashes are acceptable);
9. Patient with current alcohol abuse or actively consuming drugs (addiction); as it may interfere with patient's ability to comply with study procedures
10. Periodontal surgery planned during the study;
11. Female patient pregnant, nursing or planning to become pregnant within the next 12 months;
12. Patient is a current smoker or had been smoking or using nicotine product(s) in the last six months;
13. Concurrent disease (such as porphyria) or drug(s) (such as methotrexate or chloroquine) known to induce severe photosensitivity of the skin;
14. Patient has ongoing malignant disease of any type, or any significant chronic disease which, in the opinion of the investigator, might interfere with the evaluation of the study objectives or would result in non-compliance with the study protocol;
15. Patients with known hypersensitivity to peroxide;
16. Patients with known photosensitivity or who take drugs to treat photosensitivity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-11; Primary Completion 2015-03 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Adverse events, Serious adverse events and incidents | 3 weeks
  Number of patients with adverse events, serious adverse events and incidents
Ease of performing SRP and time required to perform SRP | 2 weeks

SECONDARY OUTCOMES:
Impact on tissues (Visual examination of tissues) | 3 weeks
  Visual examination of tissues
Impact on bleeding (Use of Bleeding on Probing (BOP) results) | 2 weeks
  Use of Bleeding on Probing (BOP) results
Impact on Plaque Index (PI) | 2 weeks
Impact on Gingival index (GI) | 2 weeks
Pain (Visual Analog Scale) | 2 weeks

OTHER OUTCOMES:
Exploratory endpoint: patient's preference questionnaire | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Seminara, DDM, Principal Investigator — Dr. Anthony Seminara Inc.
Locations (1):
- Dr. Anthony Seminara Inc., Montreal, Quebec, Canada